CLINICAL TRIAL: NCT06670248
Title: GlycoBURN Study: Determination of Endothelial Glycocalyx Status in the Surgical Resuscitation of Severe Burn Patients
Brief Title: Evaluation of Endothelial Glycocalyx in the Surgical Resuscitation of Major Burn Patients
Acronym: GlycoBURN
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AT)400/2023
Record Dates: First submitted 2024-10-23; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Syndecan 1; Severe Burn; Endotheliopathy of Trauma; Endothelial Glycocalyx; Hemorrhagic Shock; Postoperative Complications
Keywords: Syndecan 1; Endotheliopathy; Glycocalyx; Proteoglycan; Severe burn
MeSH Terms: conditions — Burns; Shock, Hemorrhagic; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All blood samples will be properly labeled with each patient's identification and sent to the central laboratory of our hospital, where they will be centrifuged and stored at -80ºC. Sample processing will be conducted once all patients have been recruited. The analysis of syndecan-1 will be performed using an enzyme-linked immunosorbent assay (ELISA). Each blood draw will consist of 10 ml. No DNA analysis will be conducted at any point; only syndecan-1 levels will be measured
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Severe burn patients: Adult severely burned patients (TBSA ≥ 20%) undergoing debridement surgery.
  Interventions: Procedure: Debridement Surgery; Diagnostic Test: Sdc-1 Level Measurement

INTERVENTIONS:
Procedure: Debridement Surgery — Surgical debridement of burn wounds involving ≥ 20% of the TBSA, including debrided and donor sites.
Diagnostic Test: Sdc-1 Level Measurement — Measurement of plasma sdc-1 levels in different situations to assess endothelial glycocalyx damage using an enzyme-linked immunosorbent assay (ELISA):
  Preoperatively:
  * Upon admission to the Burn Unit.
  * 24 hours after admission to the Burn Unit.
  * Prior to the start of surgery, after anesthetic induction.
  * If surgery is performed after the fifth day following the burn, an additional sdc-1 measurement will be taken on the fifth day of hospital admission.
  Postoperatively:
  * 6 hours after surgery.
  * 24 hours after surgery.
  * 48 hours after surgery.

SUMMARY:
The purpose of this observational study is to examine whether Endotheliopathy of Trauma (EoT) is present in severely burned patients and how it is affected by burn debridement surgery.

The main questions it aims to answer are:

* Do severely burned patients present with EoT before undergoing burn debridement surgery?
* Does the surgical intervention worsen EoT, leading to increased postoperative syndecan 1 (sdc 1) levels compared to preoperative levels?

Participants will:

* Undergo debridement surgery where the total area of debrided and donor sites covers 20% or more of the Total Body Surface Area (TBSA).
* Have their sdc 1 levels measured before and after surgery.
* Have perioperative factors analyzed to assess their impact on endothelial damage and glycocalyx functionality.

This study aims to provide insight into how surgical resuscitation affects the endothelial glycocalyx in severely burned patients.

DETAILED DESCRIPTION:
The endothelial glycocalyx is a protective layer of glycoproteins, glycosaminoglycans, and proteoglycans that lines the luminal surface of blood vessels and plays a critical role in regulating vascular permeability and coagulation. The syndecan family, consisting of four members (syndecan 1-4), is the main proteoglycan. Of particular interest, sdc 1 is a marker of endothelial damage, with elevated levels (>40 ng/ml) being linked to EoT. This condition is characterized by increased transfusion requirements, prolonged hospital stays, and higher morbidity and mortality rates.

Early burn debridement (from the fifth day onward) has been associated with improved outcomes in severely burned patients. The purpose of this surgical intervention is to mitigate the inflammatory response triggered by the burned (and potentially infected) skin. However, this surgery presents significant challenges for anesthesiologists, as it typically involves massive blood loss and may exacerbate the shock that these patients frequently experience. To counteract hemorrhagic shock induced by the surgical trauma, fluid and blood product administration is critical. The state of the endothelial glycocalyx may influence the effectiveness of surgical resuscitation. When damaged, the glycocalyx heightens the risk of postoperative pulmonary edema, prolonged mechanical ventilation, abdominal or limb compartment syndrome, and deepened burns due to poor perfusion. These complications increase the likelihood of sepsis, multi-organ failure, and elevated mortality.

This study aims to evaluate whether EoT is present in severely burned patients before surgery and assess whether the surgical intervention exacerbates this condition. Investigators will conduct a two-year prospective observational cohort study at the Burn Unit of Vall d'Hebron University Hospital, from March 2024 to March 2026. The study will include patients undergoing burn debridement surgery involving 20% or more of their TBSA. Plasma sdc 1 levels will be measured preoperatively and postoperatively to assess glycocalyx disruption. Additionally, investigators will analyze perioperative factors to determine their relationship with endothelial damage.

The literature on severely burned patients and the endothelial glycocalyx is limited, with no studies to date specifically addressing its role in surgical resuscitation. Quantifying perioperative sdc 1 levels will help provide a clearer understanding of the status and function of the glycocalyx in these patients. This insight could contribute to strategies aimed at protecting the endothelial glycocalyx, potentially reducing postoperative complications related to fluid therapy and positively impacting the morbidity and mortality of severely burned patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with burned TBSA greater than or equal to 20%.
* Patients who will undergo debridement of at least 20% of the burned TBSA (including the debrided area and the donor site).

Exclusion Criteria:

* Under 18 years old.
* Pregnant women.
* Patient refusal.
* Polytraumatized patients.
* Electrical or chemical burns.
* Patients with any of the following pre-burn conditions: complicated heart disease*, renal disease on hemodialysis/hemofiltration or with Glomerular Filtration Rate (GFR) < 30 ml/min/1.73m², and liver cirrhosis (Child A, B, and C).

(* Definition of complicated heart disease: decompensated heart failure (NYHA class IV), Left Ventricular Ejection Fractio < 40%, or severe valvular disease).

* Patients with a history of chronic inflammatory diseases (autoimmune disease).
* Patients on chronic treatment with corticosteroids or immunosuppressants.
* Patients requiring reintervention for debridement surgery who have already been included in the study during their first surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Burn Unit of Vall d'Hebron University Hospital with burned TBSA ≥ 20% who undergo debridement surgery (total area between the debrided and donor sites ≥ 20% of TBSA).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Sdc-1 perioperative changes | From admission to our Burn Unit until 48 hours post-debridement surgery.
  Sdc-1 levels will be measured upon admission to our Burn Unit, 24 hours after admission, on the 5th day of admission if surgery has not yet been performed, immediately before debridement surgery, and during the first 48 hours postoperatively.

SECONDARY OUTCOMES:
Postoperative complications | A) Immediate complications: 24 hours postoperatively; B) Early complications: 7 days postoperatively; C) Late complications: 30 days postoperatively
  1. Cardiovascular complications (yes/no): new-onset atrial fibrillation or other arrhythmias, presence of non-fatal cardiopulmonary arrest, acute myocardial infarction, acute pulmonary edema, and myocardial injury after non-cardiac surgery (MINS).
  2. Pulmonary complications (yes/no): pneumonia, whether associated with mechanical ventilation or not, pleural effusion, acute respiratory distress syndrome (ARDS), pneumothorax, bronchospasm, and the need for tracheostomy.
  3. Renal failure (yes/no): need for dialysis or hemofiltration (yes/no).
  4. Abdominal compartment syndrome (yes/no).
  5. Thrombotic complications (yes/no): lower limb thrombosis, pulmonary embolism, and cerebrovascular accident.
  (The following publication is used as a reference for the definition of complications: DOI: 10.1097/EJA.0000000000000118).
Fluid and transfusion requirements | During the surgical procedure and the first 48 hours postoperatively.
  Volume of fluids and blood products transfused during surgery and in the postoperative period.
Coagulation abnormalities (preoperative and postoperative) | Preoperative (from admission to surgery) and postoperative (up to 48 hours after surgery).
  Analysis of the coagulation abnormalities (guided by classic coagulation tests and thromboelastometry parameters) resulting from burn debridement surgery
Duration of Mechanical Ventilation | From the end of surgery until extubation, assessed over a period of up to 180 days.
  Number of days on mechanical ventilation after debridement surgery
Length of Stay in the Intensive Care Unit (ICU) | From admission to the ICU, after de debridement surgery, until discharge from the ICU (assessed over a period of up to 180 days).
  Number of days of ICU stay
Survival of severely burned patients after debridement surgery | From surgery until 180 days postoperatively.
  Survival from surgery until 180 days postoperatively.

OTHER OUTCOMES:
Inhalation injury | At admission
  Incidence of inhalation injury in severely burned patients
Preoperative complications | From admission to the Burn Unit until the day of the first debridement surgery, assessed over a period of up to 30 days following admission.
  Incidence of pre-surgical complications including: pulmonary infection, urinary tract infection, renal dysfunction, skin infection, shock, pulmonary distress, ischemic heart disease, atrial fibrillation, thrombotic or hemorrhagic stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that will be shared include:
  * Demographic data (e.g., age, sex, weight, height,)
  * Clinical data (e.g., medical history, burn characteristics, TBSA, type of burn)
  * Outcome measures (e.g., syndecan-1 levels, postoperative complications, survival rates)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and supporting information will be available starting 6 months after the final study results are published and will remain available for 5 years.
Access Criteria: Qualified researchers affiliated with academic, medical, or scientific institutions will be able to access the IPD and supporting information. They will be able to access de-identified individual participant data, including demographic information, clinical data, and outcome measures. Researchers can request access to the data by submitting a data-sharing proposal to Vall d'Hebron University Hospital and signing a data use agreement. Requests will be evaluated on a case-by-case basis.

REFERENCES:
- [Background] Keyloun JW, Le TD, Brummel-Ziedins KE, Mclawhorn MM, Bravo MC, Orfeo T, Johnson LS, Moffatt LT, Pusateri AE, Shupp JW; SYSCOT Study Group. Inhalation Injury Is Associated With Endotheliopathy and Abnormal Fibrinolytic Phenotypes in Burn Patients: A Cohort Study. J Burn Care Res. 2022 Mar 23;43(2):432-439. doi: 10.1093/jbcr/irab102. PMID 34089618
- [Background] Keyloun JW, Le TD, Pusateri AE, Ball RL, Carney BC, Orfeo T, Brummel-Ziedins KE, Bravo MC, McLawhorn MM, Moffatt LT, Shupp JW; and the SYSCOT study group. Circulating Syndecan-1 and Tissue Factor Pathway Inhibitor, Biomarkers of Endothelial Dysfunction, Predict Mortality in Burn Patients. Shock. 2021 Aug 1;56(2):237-244. doi: 10.1097/SHK.0000000000001709. PMID 33394974
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Luker JN, Vigiola Cruz M, Carney BC, Day A, Moffatt LT, Johnson LS, Shupp JW. Shedding of the endothelial glycocalyx is quantitatively proportional to burn injury severity. Ann Burns Fire Disasters. 2018 Mar 31;31(1):17-22. PMID 30174566
- [Background] Osuka A, Kusuki H, Yoneda K, Matsuura H, Matsumoto H, Ogura H, Ueyama M. Glycocalyx Shedding is Enhanced by Age and Correlates with Increased Fluid Requirement in Patients with Major Burns. Shock. 2018 Jul;50(1):60-65. doi: 10.1097/SHK.0000000000001028. PMID 29023362
- [Background] Welling H, Henriksen HH, Gonzalez-Rodriguez ER, Stensballe J, Huzar TF, Johansson PI, Wade CE. Endothelial glycocalyx shedding in patients with burns. Burns. 2020 Mar;46(2):386-393. doi: 10.1016/j.burns.2019.05.009. Epub 2019 Dec 20. PMID 31866179
- [Background] Rodriguez EG, Ostrowski SR, Cardenas JC, Baer LA, Tomasek JS, Henriksen HH, Stensballe J, Cotton BA, Holcomb JB, Johansson PI, Wade CE. Syndecan-1: A Quantitative Marker for the Endotheliopathy of Trauma. J Am Coll Surg. 2017 Sep;225(3):419-427. doi: 10.1016/j.jamcollsurg.2017.05.012. Epub 2017 Jun 1. PMID 28579548
- [Background] Johansson PI, Stensballe J, Ostrowski SR. Shock induced endotheliopathy (SHINE) in acute critical illness - a unifying pathophysiologic mechanism. Crit Care. 2017 Feb 9;21(1):25. doi: 10.1186/s13054-017-1605-5. PMID 28179016
- [Background] Tapking C, Hernekamp JF, Horter J, Kneser U, Haug V, Vogelpohl J, Schulte M, Kremer T, Hundeshagen G. Influence of burn severity on endothelial glycocalyx shedding following thermal trauma: A prospective observational study. Burns. 2021 May;47(3):621-627. doi: 10.1016/j.burns.2020.07.021. Epub 2020 Aug 5. PMID 32839038
- [Background] Abdullah S, Karim M, Legendre M, Rodriguez L, Friedman J, Cotton-Betteridge A, Drury R, Packer J, Guidry C, Duchesne J, Taghavi S, Jackson-Weaver O. Hemorrhagic Shock and Resuscitation Causes Glycocalyx Shedding and Endothelial Oxidative Stress Preferentially in the Lung and Intestinal Vasculature. Shock. 2021 Nov 1;56(5):803-812. doi: 10.1097/SHK.0000000000001764. PMID 34259440
- [Background] Bunch CM, Chang E, Moore EE, Moore HB, Kwaan HC, Miller JB, Al-Fadhl MD, Thomas AV, Zackariya N, Patel SS, Zackariya S, Haidar S, Patel B, McCurdy MT, Thomas SG, Zimmer D, Fulkerson D, Kim PY, Walsh MR, Hake D, Kedar A, Aboukhaled M, Walsh MM. SHock-INduced Endotheliopathy (SHINE): A mechanistic justification for viscoelastography-guided resuscitation of traumatic and non-traumatic shock. Front Physiol. 2023 Feb 27;14:1094845. doi: 10.3389/fphys.2023.1094845. eCollection 2023. PMID 36923287
- [Background] Basas VA, Schutzman LM, Brown IE. Implications of the Regulation of Endothelial Glycocalyx Breakdown and Reconstitution in Severe Burn Injury. J Surg Res. 2023 Jun;286:110-117. doi: 10.1016/j.jss.2022.12.033. Epub 2023 Feb 17. PMID 36804690
- [Background] Vigiola Cruz M, Carney BC, Luker JN, Monger KW, Vazquez JS, Moffatt LT, Johnson LS, Shupp JW. Plasma Ameliorates Endothelial Dysfunction in Burn Injury. J Surg Res. 2019 Jan;233:459-466. doi: 10.1016/j.jss.2018.08.027. Epub 2018 Sep 22. PMID 30502286